CLINICAL TRIAL: NCT01384149
Title: A Pioneer Study: External Selective Laser Trabeculoplasty for Treating Uncontrolled Open Angle Glaucoma
Brief Title: EXTERNAL SLT Treatment in Patients With Uncontrolled OPEN ANGLE GLAUCOMA
Acronym: ETSG
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Meir Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: meirslt2011
Record Dates: First submitted 2011-05-16; First posted 2011-06-28 (Estimated); Last update posted 2014-08-12 (Estimated); Status verified 2014-08

CONDITIONS: Primary Open Angle Glaucoma
Keywords: intra ocular pressure; open angle glaucoma; selective laser trabeculoplasty; external laser treatment
MeSH Terms: conditions — Glaucoma, Open-Angle

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- standart slt (Active Comparator): gonioscopic selective laser trabeculoplasty
  Interventions: Device: standard slt
- external slt (Experimental): perilimbal ,above trabecular meshwork 180 degrees ,100 laser dots
  Interventions: Device: external slt

INTERVENTIONS:
Device: external slt — Nd:YAG LASER SLT perilimbal above trabecular meshwork 180 degrees ,100 lasering dots
  Other Names: external SLT laser
  Arms: external slt
Device: standard slt — Nd:YAG LASER SLT gonioscopic laser treatment
  Other Names: SLT laser
  Arms: standart slt

SUMMARY:
The purpose of this study is to evaluate the advantages and disadvantages of external selective laser trabeculoplasty (SLT) in treating open angle glaucoma,compared to traditional SLT.

DETAILED DESCRIPTION:
glaucoma is the 2nd leading cause for blindness in the western world.at the time approximately 60 million people are diagnosed as glaucoma patients with an estimated rise of 30% in the next decade. glaucoma is defined as a progressive damage to the optic nerve ,followed by a damage to the visual field. high intraocular pressure (IOP) is considered a main risk factor.lowering IOP can be done in several ways ,including medication ,laser treatment and operations.

medical treatment is effective in most cases ,but requires high daily compliance,side effects and availability of medication in living areas.

laser trabeculoplasty treatment for reducing IOP is a first line treatment for patients with open angle glaucoma (OAG).with success rate of 70-90%, it can be done as an additive treatment or as a sole treatment.

SLT or "cold" laser is a non-invasive treatment in which short wave lengths are being transduced in short intervals ,through a gonioscopic lens to the area of filtering angle. thec wave length is specific to cells rich in melanin (located in the filtering angle). the mechanism of action is regeneration of cytokine surge -causing macrophages recruitment and breakage of inter-cell connections at the trabecular meshwork (filtering area) and allows rise in fluid shift. the treatment requires several lasering to areas at the surrounding the wave does not cause rise in tissue heat or scaring of tissue and can be repeated.among its disadvantages are reduction in affect during time,causing new elevation of IOP , potential peripheral anterior synechia (PAS), corneal erosion or oedema,requires experience in treating through gonioscopic lense.

previous reports in the literature regarding external low intensity laser (LIL)show less complication rate.

our study evaluates the use of external SLT by using a standard retinal laser machine ,with procedure performed on the outer sclera-above the trabecular meshwork with laser parameters similar to those used in retinal surgeries.

this is a prospective, randomized, comparative clinical trial.

ELIGIBILITY:
Inclusion Criteria:

* Primary Open Angle Glaucoma
* clinical appearance of pigment at the angle
* angle assessed as >3 by a professional glaucoma expert
* IOP above target pressure under full anti-hypertensive treatment with a good compliance for treatment or IOP above target pressure and poor compliance to medical treatment due to: allergic reaction , side effects,physical inability etc.
* able to sign independently on an informed concent

Exclusion Criteria:

* pregnancy/breast feeding
* glaucoma not specified as primary open angle glaucoma
* sensitivity to on or more of the medications in the study
* current /past intraocular inflammation
* primary open angle glaucoma with out appearance of pigment at the angle
* s/p laser trabeculoplasty at treatment eye
* inability to sign an informed concent

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2011-09; Primary Completion 2012-01 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
Intra Ocular Pressure values as a measure for treatment success | 6 months
  a success is defined a decrease of >/= 20% in intra ocular pressure measured after treatment -compared to intra ocular pressure measured prior to treatment a relative success in an intra ocular pressure thet is lowered post treatment in less than 20% -compared to pre-treatment. failure is considered as an intra ocular pressure equal or higher than measured prior to treatment

SECONDARY OUTCOMES:
Use of supplementary treatment for lowering intraocular pressure | 6 months
  success is defined as no need for suplemental medication for lowering intra ocular pressure ,complete failure is described as using the same amount or more of medication ,relative success in described as a need to use less hypotensive medications for lowering intraocular pressure after the procedure

CONTACTS AND LOCATIONS:
Overall Officials: Noa Gefen, Dr., Study Chair — Meir Medical Center, Kfar Saba, Israel; Michael Belkin, Prof., Principal Investigator — Sheba Medical Center, Ramat Gan ,Israel; Ehud Asia, Prof., Principal Investigator — Meir Medical Center, Kfar Saba, Israel; Audry masas-kaplan, Dr., Principal Investigator — Assaf Harofhe Medical Center, Beer Yaakov, Israel
Locations (3):
- Israel (3):
  - Assaf Harofhe Medical Center, Beer Yaakov
  - Ophthalmology Department ,Meir Medical Center, Kfar Saba
  - Sheba Medical Center, Ramat Gan

REFERENCES:
- [Background] Quigley HA, Broman AT. The number of people with glaucoma worldwide in 2010 and 2020. Br J Ophthalmol. 2006 Mar;90(3):262-7. doi: 10.1136/bjo.2005.081224. PMID 16488940
- [Background] The Advanced Glaucoma Intervention Study (AGIS): 7. The relationship between control of intraocular pressure and visual field deterioration.The AGIS Investigators. Am J Ophthalmol. 2000 Oct;130(4):429-40. doi: 10.1016/s0002-9394(00)00538-9. PMID 11024415
- [Background] Freeman EE, Munoz B, West SK, Jampel HD, Friedman DS. Glaucoma and quality of life: the Salisbury Eye Evaluation. Ophthalmology. 2008 Feb;115(2):233-8. doi: 10.1016/j.ophtha.2007.04.050. Epub 2007 Jul 26. PMID 17655930
- [Background] Worthen DM, Wickham MG. Argon laser trabeculotomy. Trans Am Acad Ophthalmol Otolaryngol. 1974 Mar-Apr;78(2):OP371-5. No abstract available. PMID 4856873
- [Background] Latina MA, Sibayan SA, Shin DH, Noecker RJ, Marcellino G. Q-switched 532-nm Nd:YAG laser trabeculoplasty (selective laser trabeculoplasty): a multicenter, pilot, clinical study. Ophthalmology. 1998 Nov;105(11):2082-8; discussion 2089-90. doi: 10.1016/S0161-6420(98)91129-0. PMID 9818610
- [Background] Alvarado JA, Katz LJ, Trivedi S, Shifera AS. Monocyte modulation of aqueous outflow and recruitment to the trabecular meshwork following selective laser trabeculoplasty. Arch Ophthalmol. 2010 Jun;128(6):731-7. doi: 10.1001/archophthalmol.2010.85. PMID 20547951
- [Background] Rachmiel R, Trope GE, Chipman ML, Gouws P, Buys YM. Laser trabeculoplasty trends with the introduction of new medical treatments and selective laser trabeculoplasty. J Glaucoma. 2006 Aug;15(4):306-9. doi: 10.1097/01.ijg.0000212233.11287.b3. PMID 16865007
- [Background] Coleman AL, Yu F, Evans SJ. Use of gonioscopy in medicare beneficiaries before glaucoma surgery. J Glaucoma. 2006 Dec;15(6):486-93. doi: 10.1097/01.ijg.0000212287.62798.8f. PMID 17106360
- [Background] Ivandic BT, Hoque NN, Ivandic T. Early diagnosis of ocular hypertension using a low-intensity laser irradiation test. Photomed Laser Surg. 2009 Aug;27(4):571-5. doi: 10.1089/pho.2008.2342. PMID 19514814
- [Background] Framme C, Walter A, Prahs P, Theisen-Kunde D, Brinkmann R. Comparison of threshold irradiances and online dosimetry for selective retina treatment (SRT) in patients treated with 200 nanoseconds and 1.7 microseconds laser pulses. Lasers Surg Med. 2008 Nov;40(9):616-24. doi: 10.1002/lsm.20685. PMID 18951425
- [Background] Klatt C, Saeger M, Oppermann T, Porksen E, Treumer F, Hillenkamp J, Fritzer E, Brinkmann R, Birngruber R, Roider J. Selective retina therapy for acute central serous chorioretinopathy. Br J Ophthalmol. 2011 Jan;95(1):83-8. doi: 10.1136/bjo.2009.178327. Epub 2010 Jun 15. PMID 20554506
- [Derived] Rolim-de-Moura CR, Paranhos A Jr, Loutfi M, Burton D, Wormald R, Evans JR. Laser trabeculoplasty for open-angle glaucoma and ocular hypertension. Cochrane Database Syst Rev. 2022 Aug 9;8(8):CD003919. doi: 10.1002/14651858.CD003919.pub3. PMID 35943114